CLINICAL TRIAL: NCT00492856
Title: S0521, A Randomized Trial of Maintenance Versus Observation for Patients With Previously Untreated Low and Intermediate Risk Acute Promyelocytic Leukemia (APL), Phase III
Brief Title: S0521, Combination Chemotherapy With or Without Gemtuzumab Followed By Tretinoin, Mercaptopurine, and Methotrexate or Observation in Treating Patients With Acute Promyelocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S0521; S0521 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute promyelocytic leukemia (M3); untreated adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Promyelocytic, Acute | interventions — Mercaptopurine; Methotrexate; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Post-consolidation therapy arm I (Experimental): Patients receive oral tretinoin twice daily on days 1-7, oral mercaptopurine once daily on days 1-14, and oral methotrexate on day 1. Treatment repeats every 2 weeks for up to 1 year.
  Interventions: Drug: mercaptopurine; Drug: methotrexate; Drug: tretinoin
- Post-consolidation therapy arm II (No Intervention): Patients receive no further chemotherapy. Patients are followed every 3 months for 1 year. (Randomization and observation arm closed as of 8/15/10)

INTERVENTIONS:
Drug: mercaptopurine — Given orally
  Arms: Post-consolidation therapy arm I
Drug: methotrexate — Given orally
  Arms: Post-consolidation therapy arm I
Drug: tretinoin — Given orally
  Arms: Post-consolidation therapy arm I

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as gemtuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Sometimes the cancer may not need more treatment until it progresses. In this case, observation may be sufficient. It is not yet known whether combination chemotherapy is more effective than observation when given as maintenance therapy in treating acute promyelocytic leukemia.

PURPOSE: This randomized phase III trial is studying tretinoin, mercaptopurine, and methotrexate to see how well they work when given as maintenance therapy compared with observation after combination chemotherapy in treating patients with acute promyelocytic leukemia. (Randomization and observation group closed as of 8/15/10)

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare disease-free survival (DFS) among patients with previously untreated low and intermediate risk acute promyelocytic leukemia (APL) who are PCR-negative for Promyelocytic-retinoic acid receptor alpha (PML-RARα) after consolidation therapy and receive maintenance therapy versus patients who receive no maintenance therapy. (Randomization and observation arm closed as of 8/15/10)
* Assess the toxicity of induction, consolidation and maintenance in these patients.
* Test whether gene expression profiles assessed prior to treatment are predictive of resistance to remission induction chemotherapy and correlate with detectable minimal residual disease post-consolidation therapy. (Only one patient was not in molecular remission after receiving consolidation. Therefore, the predictive value of pre-treatment gene expression profiling could not be determined and is not reported here).
* Investigate in a preliminarily manner the outcomes of patients who fail to achieve or maintain PCR-negative PML-RARα fusion gene after consolidation therapy when treated with gemtuzumab ozogamicin. (Only one patient was treated with gemtuzumab ozogamicin as part of protocol treatment. Therefore, results for this objective are not reported).

OUTLINE: This is a randomized, multicenter study.

* Induction therapy: Patients receive oral tretinoin twice daily until morphologic complete remission (CR) or for a maximum of 90 days in the absence of disease progression or unacceptable toxicity. Patients also receive cytarabine IV continuously on days 3-9 and daunorubicin hydrochloride IV on days 3-6.
* Consolidation therapy: Patients who achieve CR, CR with incomplete blood count recovery (CRi), or partial remission (PR) after induction therapy receive arsenic trioxide IV over 2 hours 5 days a week for 5 weeks. After a 2-week rest period, patients receive a second course of arsenic trioxide. Within 14-30 days after blood count recovery, patients receive oral tretinoin twice daily on days 1-7 and daunorubicin hydrochloride IV on days 1-3. Patients receive a second course of tretinoin and daunorubicin hydrochloride after adequate blood count recovery.
* Post-consolidation therapy: Patients who do not achieve molecular CR (CRm), but do achieve CR or CRi and are still PML-RARα-positive after consolidation therapy, receive gemtuzumab ozogamicin IV over 2 hours on days 1 and 15. Treatment repeats every 14 days for up to 6 courses or until PML-RARα-negative by PCR. (closed as of 8/15/10)Patients are stratified according to age (18 to 60 years vs > 60 years), acute promyelocytic leukemia (APL) risk group (low vs intermediate), and if the patient received consolidation therapy courses 3 or 4 (yes vs no) regardless of their CRm response. These patients are randomized to 1 of 2 treatment arms. (Randomization and observation arm closed as of 8/15/10) All patients are non-randomly assigned to receive post-consolidation therapy.

  * Arm I: Beginning 14-30 days after blood count recovery, patients receive oral tretinoin twice daily on days 1-7, oral mercaptopurine once daily on days 1-14, and oral methotrexate on day 1. Treatment repeats every 2 weeks for up to 1 year.
  * Arm II: Patients receive no further chemotherapy. Patients are followed every 3 months for 1 year. (Randomization and observation arm closed as of 8/15/10) Patients undergo blood collection periodically for cytogenetic studies. Samples are analyzed for PML-RARα fusion gene via reverse transcriptase-polymerase chain reaction (RT-PCR) assay and gene expression profiling.

After completion of study treatment, patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically confirmed acute promyelocytic leukemia (APL) or the variant form of APL

  * Previously untreated disease
  * Low- or intermediate-risk disease

    * Low-risk disease, defined as white blood cell (WBC) ≤ 10,000/mm^3 and platelet count > 40,000/mm^3
    * Intermediate-risk disease, defined as WBC ≤ 10,000/mm^3 and platelet count ≤ 40,000/mm^3
    * WBC and platelet count confirming low- or intermediate-risk disease must be obtained within 48 hours prior to study registration unless the patient received tretinoin therapy prior to study registration in which case the WBC and platelet count must be obtained within 48 hours prior to study therapy
* PML-RARα fusion gene positive by reverse transcriptase-polymerase chain reaction (RT-PCR) assay
* No recurrent disease
* Must be registered on clinical trials SWOG-9007 and SWOG-S9910

  * Specimens must be collected prior to tretinoin therapy and may be collected after tretinoin therapy

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-3
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for ≥ 1 month prior to, during, and for 2 months after completion of study treatment
* No unstable cardiac arrhythmia or unstable angina
* No other malignancy within the past 5 years except for the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * Carcinoma in situ of the cervix
  * Adequately treated stage I or II cancer (except for highly aggressive malignancies with a high rate of early relapse) currently in complete remission

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than 1 prior dose of intrathecal chemotherapy for acute leukemia
* No prior systemic chemotherapy, hydroxyurea, or leukapheresis for acute leukemia

  * Prior tretinoin at a dose of ≤ 45 mg/m^2/day allowed provided it was received ≤ 5 days prior to study registration

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2007-06-01; Primary Completion 2013-12-01 (Actual); Study Completion 2016-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven E. Coutre, MD, Study Chair — Stanford University
Locations (210):
- United States (210):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - Stanford Cancer Center, Stanford, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Hematology Oncology Associates of Illinois - Berwyn, Berwyn, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Kellogg Cancer Care Center, Highland Park, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - La Grange Oncology Associates - Geneva, Naperville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Derived] Coutre SE, Othus M, Powell B, Willman CL, Stock W, Paietta E, Levitan D, Wetzler M, Attar EC, Altman JK, Gore SD, Maher T, Kopecky KJ, Tallman MS, Larson RA, Appelbaum FR. Arsenic trioxide during consolidation for patients with previously untreated low/intermediate risk acute promyelocytic leukaemia may eliminate the need for maintenance therapy. Br J Haematol. 2014 May;165(4):497-503. doi: 10.1111/bjh.12775. Epub 2014 Feb 14. PMID 24528179

RESULTS

PARTICIPANT FLOW:
Groups:
- Low and Intermediate Risk APL Patients: All patients received induction: ATRA 45 mg/m^2/day orally, divided BID, Ara-C 200 mg/m^2/day continuous IV infusion days 3-9, Daunorubicin 50 mg/m^2/day IV bolus days 3-6. If CR (CRm), CRi, or PR, patients received consolidation: Arsenic trioxide 0.15 mg/kg/day IV infusion over 2 hours, 5 days per week for 5 weeks followed by 2 weeks of rest (2 courses). ATRA 45 mg/m^2/day orally divided BID days 1-7, Daunorubicin 50 mg/m^2/day IV bolus days 1-3 (2 courses).
- Post-consolidation ATRA, 6-MP, MTX: Patients who achieved CRm after consolidation and were randomized or assigned to the treatment arm received ATRA 45 mg/m^2/day orally divided BID 7 days repeated every other week, 6-MP 60 mg/m^2/day orally daily, Methotrexate 20 mg/m^2 orally once a week (1 year cycle). Effective with Revision #6, all eligible patients were non-randomly assigned to receive maintenance with ATRA, 6-MP, and MTX.
- Post-consolidation Observation: Patients who achieved CRm after consolidation and were randomized to the observation arm.
- Post-consolidation Gemtuzumab Ozogamicin: Patients who did not achieve CRm, but achieved CR/CRi and are PML-RARα-positive after consolidation received maintenance gemtuzumab ozogamicin 6 mg/m^2/day IV over 2 hours days 1 and 15 (up to 6 does).
Period: Induction
Arm/Group | Low and Intermediate Risk APL Patients | Post-consolidation ATRA, 6-MP, MTX | Post-consolidation Observation | Post-consolidation Gemtuzumab Ozogamicin
Started | 105 | 0 | 0 | 0
Completed | 99 | 0 | 0 | 0
Not Completed | 6 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Death | 3 | 0 | 0 | 0
Period: Consolidation
Arm/Group | Low and Intermediate Risk APL Patients | Post-consolidation ATRA, 6-MP, MTX | Post-consolidation Observation | Post-consolidation Gemtuzumab Ozogamicin
Started | 92 (Patients in CR (CRm), CRi, or PR after induction, register for consolidation and are eligible.) | 0 | 0 | 0
Completed | 83 | 0 | 0 | 0
Not Completed | 9 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 0 | 0 | 0
Not completed — Not protocol specified | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Period: Post-consolidation
Arm/Group | Low and Intermediate Risk APL Patients | Post-consolidation ATRA, 6-MP, MTX | Post-consolidation Observation | Post-consolidation Gemtuzumab Ozogamicin
Started | 0 (Patients who achieve CRm, are randomized to the treatment arm, and are eligible.) | 41 | 27 | 1
Completed | 0 | 29 | 0 | 0
Not Completed | 0 | 12 | 27 | 1
Not completed — Adverse Event | 0 | 4 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Not protocol specified | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0
Not completed — Observation Arm | 0 | 0 | 27 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low and Intermediate Risk APL Patients: All patients received induction: ATRA 45 mg/m^2/day orally, divided BID, Ara-C 200 mg/m^2/day continuous IV infusion days 3-9, Daunorubicin 50 mg/m^2/day IV bolus days 3-6. If CR (CRm), CRi, or PR, patients received consolidation: Arsenic trioxide 0.15 mg/kg/day IV infusion over 2 hours, 5 days per week for 5 weeks followed by 2 weeks of rest (2 courses). ATRA 45 mg/m^2/day orally divided BID days 1-7, Daunorubicin 50 mg/m^2/day IV bolus days 1-3 (2 courses). If CRm, patients randomized to either (1) maintenance: ATRA 45 mg/m^2/day orally divided BID 7 days repeated every other week, 6-MP 60 mg/m^2/day orally daily, Methotrexate 20 mg/m^2 orally once a week (1 year cycle), or (2) observation. If CR or CRi, but not CRm, patients received maintenance gemtuzumab ozogamicin 6 mg/m^2/day IV over 2 hours days 1 and 15 (up to 6 does). Effective with Revision #6, all eligible patients were non-randomly assigned to receive maintenance with ATRA, 6-MP, and MTX.
Arm/Group | Low and Intermediate Risk APL Patients
Number analyzed (Participants) | 105
Age, Continuous [Median (Full Range); unit: years] | 49 [21 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 87
  More than one race | 0
  Unknown or Not Reported | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 87
  Unknown or Not Reported | 12

OUTCOME MEASURES:

1. Secondary Outcome: Number of Patients With Grade 3 Through 5 Adverse Events That Are Related to Study Drug
Description: Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which were deemed to be related to protocol treatment are included. Only adverse events that are possibly, probably, or definitely related to study drug are reported.
Time Frame: Up to 5 years
Population: Eligible patients who received any treatment and were assessed for adverse events were included in the adverse event summaries.
Measure: Number; unit: Participants
Groups:
- ATRA + Ara-C + Daunorubicin: ATRA 45 mg/m^2/day orally, divided BID, Ara-C 200 mg/m^2/day continuous IV infusion days 3-9, Daunorubicin 50 mg/m^2/day IV bolus days 3-6
- Consolidation: Arsenic trioxide 0.15 mg/kg/day IV infusion over 2 hours, 5 days per week for 5 weeks followed by 2 weeks of rest (2 courses). ATRA 45 mg/m^2/day orally divided BID days 1-7, Daunorubicin 50 mg/m^2/day IV bolus days 1-3 (2 courses).
- ATRA+6-MP+MTX: ATRA 45 mg/m^2/day orally divided BID 7 days repeated every other week, 6-MP 60 mg/m^2/day orally daily, Methotrexate 20 mg/m^2 orally once a week (1 year cycle).
- Gemtuzumab Ozogamicin: Gemtuzumab Ozogamicin 6 mg/m^2/day IV over 2 hours days 1 and 15 (up to 6 does)
Arm/Group | ATRA + Ara-C + Daunorubicin | Consolidation | ATRA+6-MP+MTX | Gemtuzumab Ozogamicin
Number analyzed (Participants) | 105 | 90 | 38 | 1
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 5 | 3 | 2 | 0
  AST, SGOT | 2 | 2 | 1 | 0
  Acidosis (metabolic or respiratory) | 1 | 0 | 0 | 0
  Albumin, serum-low (hypoalbuminemia) | 4 | 0 | 0 | 0
  Alkaline phosphatase | 1 | 0 | 0 | 0
  Alkalosis (metabolic or respiratory) | 2 | 0 | 0 | 0
  Anorexia | 4 | 1 | 0 | 0
  Bilirubin (hyperbilirubinemia) | 7 | 0 | 1 | 0
  CPK (creatine phosphokinase) | 2 | 0 | 0 | 0
  Calcium, serum-low (hypocalcemia) | 3 | 1 | 0 | 0
  Cardiac Arrhythmia-Other (Specify) | 1 | 0 | 0 | 0
  Cardiac troponin T (cTnT) | 2 | 0 | 0 | 0
  Cholesterol, serum-high (hypercholesterolemia) | 1 | 0 | 0 | 0
  Coagulation-Other (Specify) | 2 | 0 | 0 | 0
  Confusion | 4 | 0 | 0 | 0
  Creatinine | 2 | 0 | 0 | 0
  DIC (disseminated intravascular coagulation) | 11 | 0 | 0 | 0
  Dehydration | 0 | 1 | 0 | 0
  Diarrhea | 11 | 0 | 0 | 0
  Distention/bloating, abdominal | 2 | 0 | 0 | 0
  Dizziness | 1 | 0 | 0 | 0
  Dry skin | 1 | 0 | 0 | 0
  Dysphagia (difficulty swallowing) | 0 | 1 | 0 | 0
  Dyspnea (shortness of breath) | 11 | 0 | 0 | 0
  Enteritis (inflammation of the small bowel) | 1 | 0 | 0 | 0
  Extremity-lower (gait/walking) | 1 | 0 | 0 | 0
  Fatigue (asthenia, lethargy, malaise) | 8 | 5 | 1 | 0
  Febrile neutropenia | 58 | 8 | 0 | 1
  Fever in absence of neutropenia, ANC lt1.0x10e9/L | 1 | 1 | 0 | 0
  Flu-like syndrome | 0 | 1 | 0 | 0
  Glucose, serum-high (hyperglycemia) | 4 | 5 | 0 | 0
  Hemoglobin | 37 | 4 | 3 | 0
  Hemorrhage, CNS | 1 | 0 | 0 | 0
  Hemorrhage, GI - Rectum | 1 | 0 | 0 | 0
  Hemorrhage, GU - Vagina | 1 | 0 | 0 | 0
  Hemorrhage, pulmonary/upper respiratory - Lung | 1 | 0 | 0 | 0
  Hemorrhage, pulmonary/upper respiratory - Nose | 2 | 0 | 0 | 0
  Hypertension | 3 | 1 | 0 | 0
  Hypotension | 1 | 2 | 0 | 0
  Hypoxia | 6 | 0 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 10 | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Cecum | 1 | 0 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Colon | 4 | 0 | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Dental-tooth | 1 | 0 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 8 | 0 | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Oral cav-gums | 1 | 0 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Sinus | 0 | 0 | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Skin | 3 | 0 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - UTI | 1 | 0 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Up aerodigest | 1 | 0 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Bladder | 0 | 0 | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Blood | 1 | 5 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Catheter | 0 | 1 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Gallbladd | 1 | 0 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Skin | 3 | 1 | 0 | 0
  Inf w/unknown ANC - Oral cavity-gums (gingivitis) | 1 | 0 | 0 | 0
  Infection with unknown ANC - Bladder (urinary) | 1 | 0 | 0 | 0
  Infection with unknown ANC - Lung (pneumonia) | 1 | 0 | 0 | 0
  Infection with unknown ANC - Rectum | 1 | 0 | 0 | 0
  Infection with unknown ANC - Skin (cellulitis) | 1 | 0 | 0 | 0
  Infection-Other (Specify) | 2 | 0 | 0 | 0
  Left ventricular systolic dysfunction | 0 | 3 | 3 | 0
  Leukocytes (total WBC) | 34 | 37 | 3 | 0
  Lymphopenia | 20 | 20 | 7 | 0
  Metabolic/Laboratory-Other (Specify) | 1 | 0 | 0 | 0
  Mood alteration - agitation | 1 | 0 | 0 | 0
  Mood alteration - anxiety | 0 | 1 | 0 | 0
  Mood alteration - depression | 1 | 0 | 0 | 0
  Mucositis/stomatitis (clinical exam) - Oral cavity | 3 | 0 | 1 | 0
  Mucositis/stomatitis (clinical exam) - Rectum | 1 | 0 | 0 | 0
  Mucositis/stomatitis (functional/symp) - Oral cav | 0 | 1 | 0 | 0
  Muscle weakness, not d/t neuropathy - Extrem-lower | 1 | 0 | 0 | 0
  Muscle weakness, not d/t neuropathy - Extrem-upper | 1 | 0 | 0 | 0
  Muscle weakness, not d/t neuropathy - body/general | 2 | 0 | 0 | 0
  Myositis (inflammation/damage of muscle) | 2 | 0 | 0 | 0
  Nausea | 6 | 4 | 1 | 0
  Neuropathy: motor | 1 | 0 | 0 | 0
  Neuropathy: sensory | 0 | 2 | 0 | 0
  Neutrophils/granulocytes (ANC/AGC) | 34 | 55 | 4 | 0
  Opportunistic inf associated w/gt=Gr 2 lymphopenia | 0 | 1 | 0 | 0
  Pain - Abdomen NOS | 3 | 1 | 0 | 0
  Pain - Back | 2 | 0 | 0 | 0
  Pain - Chest/thorax NOS | 0 | 2 | 0 | 0
  Pain - Extremity-limb | 1 | 1 | 0 | 0
  Pain - Head/headache | 10 | 3 | 6 | 0
  Pain - Joint | 0 | 4 | 0 | 0
  Pain - Muscle | 3 | 2 | 0 | 0
  Pain - Neck | 1 | 0 | 0 | 0
  Pain - Rectum | 0 | 1 | 0 | 0
  Pain - Scrotum | 1 | 0 | 0 | 0
  Pain - Throat/pharynx/larynx | 0 | 1 | 0 | 0
  Pericardial effusion (non-malignant) | 1 | 1 | 0 | 0
  Pericarditis | 0 | 1 | 0 | 0
  Petechiae/purpura (hemorrhage into skin or mucosa) | 2 | 0 | 0 | 0
  Phosphate, serum-low (hypophosphatemia) | 7 | 1 | 0 | 0
  Photosensitivity | 1 | 0 | 0 | 0
  Platelets | 42 | 18 | 2 | 0
  Pleural effusion (non-malignant) | 1 | 0 | 0 | 0
  Pneumonitis/pulmonary infiltrates | 0 | 1 | 0 | 0
  Potassium, serum-low (hypokalemia) | 4 | 0 | 0 | 0
  Prolonged QTc interval | 3 | 6 | 0 | 0
  Pruritus/itching | 0 | 0 | 1 | 0
  Rash/desquamation | 3 | 1 | 0 | 0
  Renal failure | 7 | 1 | 0 | 0
  Renal/Genitourinary-Other (Specify) | 1 | 0 | 0 | 0
  Restrictive cardiomyopathy | 0 | 1 | 0 | 0
  Retinal detachment | 1 | 0 | 0 | 0
  Retinoic acid syndrome | 13 | 0 | 0 | 0
  Sodium, serum-low (hyponatremia) | 4 | 0 | 0 | 0
  Syncope (fainting) | 3 | 0 | 0 | 0
  Thrombosis/thrombus/embolism | 1 | 0 | 0 | 0
  Triglyceride, serum-high (hypertriglyceridemia) | 5 | 2 | 3 | 0
  Typhlitis (cecal inflammation) | 3 | 0 | 0 | 0
  Uric acid, serum-high (hyperuricemia) | 0 | 1 | 0 | 0
  Vasovagal episode | 1 | 1 | 0 | 0
  Ventricular arrhythmia - Ventricular tachycardia | 1 | 1 | 0 | 0
  Vomiting | 1 | 1 | 0 | 0
  Weight gain | 1 | 0 | 0 | 0

2. Primary Outcome: 3-year Disease-free Survival (DFS) Rate
Description: DFS measured from date of post-consolidation randomization until relapse of any kind or death from any cause. Observation censored at date of last follow-up for patients last known to be alive without report of relapse. Relapse from CR/CRi is occurrence of marrow blasts ≥ 5% or presence of Auer rods or presence of neoplastic promyelocytes; (re)appearance of leukemic blasts or neoplastic promyelocytes in the peripheral blood; or (re)appearance of extramedullary disease. Relapse from PR is sum of marrow blasts and promyelocytes ≥ 20%, or sum of marrow blasts and promyelocytes 6-19% with Auer rods and/or neoplastic promyelocytes; or (re)appearance of leukemic blasts or neoplastic promyelocytes in the peripheral blood; or (re)appearance of extramedullary disease. Relapse from CRc is reappearance of t(15;17) in cytogenetic analysis. Relapse from CRm/PRm is reappearance of PML-RARα by RT-PCR as defined by a normalized quotient > 10^-5 based on RT-PCR performed at appropriate central lab.
Time Frame: Up to 3 years
Population: Eligible patients in molecular remission after receiving consolidation and randomized to either maintenance chemotherapy or observation. As of 8/15/10, all eligible patients were non-randomly assigned to receive maintenance chemotherapy. Only those that were randomized to either maintenance treatment or observation were included.
Measure: Number; unit: percentage of patients
Groups:
- Post-consolidation Therapy Arm II: Patients receive no further chemotherapy. (Randomization and observation arm closed as of 05/27/10)
Arm/Group | Post-consolidation Therapy Arm I | Post-consolidation Therapy Arm II
Number analyzed (Participants) | 28 | 27
percentage of patients | 96 [90 to 100] | 100

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Eligible patients who received any treatment and were assessed for adverse events were included in the adverse event summaries.
Arm/Group | ATRA + Ara-C + Daunorubicin | Consolidation | ATRA+6-MP+MTX | Gemtuzumab Ozogamicin
Serious Adverse Events (participants affected / at risk) | 8/105 | 4/90 | 1/38 | 0/1
Other Adverse Events (participants affected / at risk) | 105/105 | 89/90 | 37/38 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATRA + Ara-C + Daunorubicin (N=105) | Consolidation (N=90) | ATRA+6-MP+MTX (N=38) | Gemtuzumab Ozogamicin (N=1)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 | 1 | 0 | 0
SVT and nodal arrhythmia - Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Extremity-lower (gait/walking) (General disorders) | 1 | 0 | 0 | 0
Sudden death (General disorders) | 1 | 1 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 1 | 0 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 0 | 1 | 0 | 0
Infection-Other (Infections and infestations) | 0 | 0 | 1 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 | 0 | 1 | 0
AST, SGOT (Investigations) | 0 | 0 | 1 | 0
Amylase (Investigations) | 0 | 0 | 1 | 0
CPK (creatine phosphokinase) (Investigations) | 1 | 0 | 0 | 0
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myositis (inflammation/damage of muscle) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATRA + Ara-C + Daunorubicin (N=105) | Consolidation (N=90) | ATRA+6-MP+MTX (N=38) | Gemtuzumab Ozogamicin (N=1)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 24 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 62 | 8 | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 43 | 59 | 22 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 4 | 7 | 3 | 0
SVT and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 3 | 2 | 2 | 0
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 13 | 10 | 0 | 0
Ventricular arrhythmia - Ventricular tachycardia (Cardiac disorders) | 5 | 6 | 0 | 0
Ocular/Visual-Other (Eye disorders) | 4 | 5 | 1 | 0
Vision-blurred vision (Eye disorders) | 6 | 7 | 2 | 0
Vision-photophobia (Eye disorders) | 0 | 0 | 2 | 0
Watery eye (epiphora, tearing) (Eye disorders) | 1 | 5 | 0 | 0
Chelitis (Gastrointestinal disorders) | 5 | 0 | 3 | 0
Constipation (Gastrointestinal disorders) | 20 | 22 | 4 | 0
Diarrhea (Gastrointestinal disorders) | 77 | 35 | 11 | 0
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 6 | 4 | 2 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 11 | 6 | 3 | 0
Hemorrhage, GI - Oral cavity (Gastrointestinal disorders) | 6 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 38 | 14 | 4 | 0
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 9 | 2 | 2 | 0
Nausea (Gastrointestinal disorders) | 72 | 66 | 26 | 0
Pain - Abdomen NOS (Gastrointestinal disorders) | 21 | 7 | 3 | 1
Vomiting (Gastrointestinal disorders) | 42 | 29 | 6 | 0
Edema: limb (General disorders) | 25 | 13 | 4 | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 67 | 70 | 27 | 1
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 29 | 16 | 3 | 0
Pain - Chest/thorax NOS (General disorders) | 8 | 16 | 4 | 0
Pain-Other (General disorders) | 5 | 3 | 1 | 1
Rigors/chills (General disorders) | 31 | 13 | 1 | 0
Allergic reaction/hypersensitivity (Immune system disorders) | 12 | 2 | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 12 | 1 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Colon (Infections and infestations) | 6 | 0 | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 15 | 2 | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 4 | 10 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 3 | 3 | 2 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Pharynx (Infections and infestations) | 0 | 2 | 2 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 6 | 6 | 2 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Up airway (Infections and infestations) | 0 | 2 | 3 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Vagina (Infections and infestations) | 0 | 1 | 2 | 0
Inf w/unknown ANC - Oral cavity-gums (gingivitis) (Infections and infestations) | 1 | 0 | 0 | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 47 | 46 | 19 | 0
AST, SGOT (Investigations) | 54 | 43 | 19 | 0
Alkaline phosphatase (Investigations) | 17 | 27 | 5 | 0
Bilirubin (hyperbilirubinemia) (Investigations) | 37 | 14 | 8 | 0
Cholesterol, serum-high (hypercholesterolemia) (Investigations) | 18 | 22 | 11 | 0
Creatinine (Investigations) | 19 | 13 | 2 | 0
Fibrinogen (Investigations) | 6 | 0 | 0 | 0
INR (of prothrombin time) (Investigations) | 11 | 1 | 4 | 0
Leukocytes (total WBC) (Investigations) | 35 | 46 | 16 | 0
Lymphopenia (Investigations) | 21 | 28 | 13 | 0
Metabolic/Laboratory-Other (Investigations) | 14 | 15 | 4 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 36 | 61 | 10 | 0
PTT (Partial thromboplastin time) (Investigations) | 16 | 6 | 4 | 0
Platelets (Investigations) | 44 | 54 | 11 | 0
Prolonged QTc interval (Investigations) | 10 | 28 | 0 | 0
Weight gain (Investigations) | 5 | 6 | 4 | 0
Weight loss (Investigations) | 15 | 6 | 1 | 0
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 37 | 19 | 6 | 0
Anorexia (Metabolism and nutrition disorders) | 45 | 16 | 5 | 0
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 7 | 5 | 1 | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 33 | 20 | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 5 | 0 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 36 | 40 | 15 | 0
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 5 | 10 | 1 | 0
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 12 | 4 | 1 | 0
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 17 | 16 | 6 | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 16 | 4 | 0 | 0
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3 | 5 | 2 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 37 | 19 | 4 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 30 | 15 | 6 | 0
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 46 | 30 | 18 | 0
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 4 | 7 | 1 | 0
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 5 | 6 | 1 | 0
Pain - Back (Musculoskeletal and connective tissue disorders) | 10 | 15 | 3 | 0
Pain - Bone (Musculoskeletal and connective tissue disorders) | 4 | 3 | 2 | 0
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2 | 0
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 12 | 10 | 3 | 0
Pain - Joint (Musculoskeletal and connective tissue disorders) | 5 | 20 | 6 | 0
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 17 | 17 | 7 | 0
Pain - Neck (Musculoskeletal and connective tissue disorders) | 7 | 3 | 1 | 0
Ataxia (incoordination) (Nervous system disorders) | 0 | 1 | 2 | 0
Dizziness (Nervous system disorders) | 12 | 21 | 6 | 0
Hemorrhage, CNS (Nervous system disorders) | 7 | 0 | 0 | 0
Neuropathy: sensory (Nervous system disorders) | 5 | 35 | 4 | 0
Ocular/Visual-Other (Nervous system disorders) | 4 | 5 | 1 | 0
Pain - Head/headache (Nervous system disorders) | 60 | 54 | 20 | 0
Taste alteration (dysgeusia) (Nervous system disorders) | 4 | 10 | 3 | 0
Tremor (Nervous system disorders) | 2 | 5 | 1 | 0
Confusion (Psychiatric disorders) | 14 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 18 | 17 | 6 | 1
Mood alteration - anxiety (Psychiatric disorders) | 15 | 11 | 5 | 0
Mood alteration - depression (Psychiatric disorders) | 14 | 4 | 4 | 0
Renal failure (Renal and urinary disorders) | 8 | 1 | 0 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 4 | 8 | 2 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 18 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 24 | 11 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 39 | 22 | 6 | 0
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 0 | 0
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 16 | 1 | 4 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 11 | 0 | 0 | 0
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 2 | 11 | 3 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 11 | 3 | 0 | 0
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 1 | 0
Retinoic acid syndrome (Respiratory, thoracic and mediastinal disorders) | 24 | 0 | 0 | 0
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 7 | 12 | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 20 | 23 | 10 | 0
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 36 | 28 | 5 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 6 | 2 | 0
Petechiae/purpura (hemorrhage into skin or mucosa) (Skin and subcutaneous tissue disorders) | 15 | 1 | 0 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 22 | 15 | 5 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 53 | 32 | 12 | 0
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 16 | 5 | 3 | 0
Hemorrhage/Bleeding-Other (Vascular disorders) | 6 | 2 | 1 | 0
Hypertension (Vascular disorders) | 21 | 5 | 3 | 0
Hypotension (Vascular disorders) | 14 | 6 | 2 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 9 | 5 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No